CLINICAL TRIAL: NCT01809977
Title: Study of Surgical Methods for Keratoconus
Brief Title: Comparison of Partial Removal and Total Removal of the Corneal Epithelium on Keratoconus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Shemshaki, MD, Research Assistant, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASD-1213-39
Record Dates: First submitted 2013-03-08; First posted 2013-03-13 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Keratoconus
Keywords: Keratoconus; remove; cornea; visual acuity
MeSH Terms: conditions — Keratoconus; Corneal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- total removal (Other): patients underwent Corneal collagen cross-linking procedure with totally corneal epithelium removing. Total removal was performed by mechanical debridement of the corneal epithelium over the central 9 mm.
  Interventions: Procedure: collagen cross-linking procedure (total removal)
- partial removal (Other): patients underwent Corneal collagen cross-linking procedure with partially corneal epithelium removing. Partial removal was performed by removing a 3-mm width ring and leaving the central 3 mm of the cornea intact.
  Interventions: Procedure: collagen cross-linking procedure (partial removal)

INTERVENTIONS:
Procedure: collagen cross-linking procedure (total removal) — patients underwent Corneal collagen cross-linking procedure with totally corneal epithelium removing. Total removal was performed by mechanical debridement of the corneal epithelium over the central 9 mm.
  Arms: total removal
Procedure: collagen cross-linking procedure (partial removal) — patients underwent Corneal collagen cross-linking procedure with partially corneal epithelium removing. Partial removal was performed by removing a 3-mm width ring and leaving the central 3 mm of the cornea intact.
  Arms: partial removal

SUMMARY:
The purpose of this study is to determine which surgical method makes less corneal haze

DETAILED DESCRIPTION:
Keratoconus is an asymmetric, bilateral, progressive non-inflammatory ectasia of the cornea. The investigators evaluate whether partial removal versus total removal of the corneal epithelium can lead to less corneal haze and better visual outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 16-40 years
* axial topography consistent with keratoconus
* minimum corneal thickness more than 400 µm and a progression of keratoconus in past 12 months

Exclusion Criteria:

* history of ocular herpes or non-healing corneal ulcers
* subjects with current ocular infection
* severe preoperative corneal haze or scar
* severe ocular surface disease
* autoimmune diseases
* pregnant women

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | at six months after surgery
  determining corrected visual acuity in partial removal versus total removal of the corneal epithelium

SECONDARY OUTCOMES:
Corneal optical density | at six months after surgery
  Corneal optical density was assessed by Scheimpflug densitometry

CONTACTS AND LOCATIONS:
Overall Officials: Behrooz Rahimi, MD, Principal Investigator — MD, Departement of ophtalmology, Isfahan University of Medical Sciences, Isfahan, Iran
Locations (1):
- Feyz university hospital, Isfahan, Isfahan, Iran

REFERENCES:
- [Derived] Razmjoo H, Rahimi B, Kharraji M, Koosha N, Peyman A. Corneal haze and visual outcome after collagen crosslinking for keratoconus: A comparison between total epithelium off and partial epithelial removal methods. Adv Biomed Res. 2014 Nov 29;3:221. doi: 10.4103/2277-9175.145677. eCollection 2014. PMID 25538907